CLINICAL TRIAL: NCT01985607
Title: Evaluation of the Efficacy of a New Thickened Extensively Hydrolyzed Formula in Infants With Cow's Milk Hypersensitivity
Brief Title: Efficacy of a New Thickened Extensively Hydrolyzed Formula
Acronym: ALLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP08-ALLAR
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Protein Allergy; Cow's Milk Protein Hypersensitivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thickened (Experimental)
  Interventions: Dietary Supplement: new extensively hydrolysed formula
- Control (Active Comparator)
  Interventions: Dietary Supplement: Extensively hydrolysed formula

INTERVENTIONS:
Dietary Supplement: new extensively hydrolysed formula
  Arms: Thickened
Dietary Supplement: Extensively hydrolysed formula
  Arms: Control

SUMMARY:
Cow Milk Allergy (CMA) occurs in 2 to 5 % of all infants. Reflux, regurgitation and vomiting are well recognised symptoms of CMA. The recommended treatment of CMA is an extensive hydrolysate. The North American Society of Pediatric Gastroenterology Hepatology and Nutrition (NASPGHAN) & the European Society of Pediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) reflux guidelines have no strict recommendations for the treatment of distressed infants with reflux, suspected of CMA. One of the preferred proposed options is to thicken an extensive hydrolysate .

This study aims at evaluating the additional value of a thickened extensive hydrolysate in children suspected of CMA and presenting with frequent regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* term born infants
* Having a Vandenplas' score of regurgitation of at least 2
* With suspected diagnosis of CMA because of clinical history/symptoms (based on a Cow's Milk Protein hypersensitivity (CMPH) score of 10 or more) and/or positive Immunoglobulin E (IgE) testing, radioallergosorbent test (RAST) or skin prick test

Exclusion Criteria:

* Exclusively breast fed infants
* Fed with an extensively hydrolysed formula or amino acid formula

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of patient dropped out for intolerance | 1 month
Vandenplas' regurgitations score | 1 month

SECONDARY OUTCOMES:
Cow's milk protein hypersensitivity score | 1 month
Growth (weight, height, head circumference) | 1 month
Growth (weight, height, head circumference) | 3 months
Growth (weight, height, head circumference) | 6 months
Number of daily regurgitations | 1 month

CONTACTS AND LOCATIONS:
Locations (5):
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Hippocration Hospital, Thessaloniki, Greece
- Faculty of Medicine, Kuwait university, Safat, Kuwait
- Pediatricians, Beirut, Lebanon
- University Children's Hospital, Ljubljana, Slovenia